CLINICAL TRIAL: NCT01272102
Title: Macular Ganglion Cell Analysis (GCA) of the Cirrus HD-OCT in Glaucoma
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: DataMed Devices Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-OCT-GCA-2010-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma: subjects with glaucoma

SUMMARY:
To determine the area under the Receiver Operator Characteristic Curve (AUC) for the Ganglion Cell Analysis (GCA) average thickness.

DETAILED DESCRIPTION:
To determine the area under the Receiver Operator Characteristic Curve (AUC) for the following GCA parameters:

1. Minimum thickness
2. Supero-temporal thickness
3. Superior thickness
4. Supero-nasal thickness
5. Infero-temporal thickness
6. Inferior thickness
7. Infero-nasal thickness

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 years or older
* Diagnosed to have glaucoma by the Principal Investigator or co-investigator
* Able and willing to make the required study visits
* Able and willing to give consent and follow study instructions

Exclusion Criteria:

Ophthalmic:

* Best corrected visual acuity in either eye worse than 20/40 on a Snellen chart or on a Snellen equivalent acuity chart.
* Refractive error outside -12.00D to +8.00D spherical range or >-3.00D cylinder.
* Previous vitreoretinal surgery in study eye.
* Vitreoretinal traction or epiretinal membrane in the study eye.
* Any active infection of anterior or posterior segments.
* Evidence of diabetic retinopathy, diabetic macular edema, or other vitreoretinal disease in the study eye upon dilated examination, or upon evaluation of retinal photos.

Systemic:

* History of diabetes, leukemia, AIDS, uncontrolled systemic hypertension, dementia or multiple sclerosis.
* A life threatening or debilitating disease.
* Participation in any study involving a non-FDA approved investigational drug (IND) within the past month, or ongoing participation in a study with a non-FDA approved or cleared investigational device (IDE).
* Current or recent (within the past 14 days) use of an agent with photosensitizing properties by any route (e.g., Visudyne®, ciprofloxacin, Bactrim®, doxycycline, etc.).
* Concomitant use of hydrochloroquine and/or chloroquine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine the area under the Receiver Operator Characteristic Curve (AUC) for the GCA average thickness, and 7 more GCA parameters. | Study was released before December 1, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Donald Budenz, MD, Principal Investigator — Bascom Palmer Eye Institute; Robert Chang, MD, Principal Investigator — Stanford Eye Institute; Arvind Neelakantan, MD, Principal Investigator — Glaucoma Associates of Texas; Alan Crandall, MD, Principal Investigator — Utah Eye Institute
Locations (4):
- United States (4):
  - Stanford Eye Institute, Palo Alto, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Glaucoma Associates of Texas, Dallas, Texas
  - Utah Eye Institute, Salt Lake City, Utah

REFERENCES:
- [Background] Tan O, Chopra V, Lu AT, Schuman JS, Ishikawa H, Wollstein G, Varma R, Huang D. Detection of macular ganglion cell loss in glaucoma by Fourier-domain optical coherence tomography. Ophthalmology. 2009 Dec;116(12):2305-14.e1-2. doi: 10.1016/j.ophtha.2009.05.025. Epub 2009 Sep 10. PMID 19744726
- [Background] Wang M, Hood DC, Cho JS, Ghadiali Q, De Moraes CG, Zhang X, Ritch R, Liebmann JM. Measurement of local retinal ganglion cell layer thickness in patients with glaucoma using frequency-domain optical coherence tomography. Arch Ophthalmol. 2009 Jul;127(7):875-81. doi: 10.1001/archophthalmol.2009.145. PMID 19597108
- [Background] Zeimer R, Asrani S, Zou S, Quigley H, Jampel H. Quantitative detection of glaucomatous damage at the posterior pole by retinal thickness mapping. A pilot study. Ophthalmology. 1998 Feb;105(2):224-31. doi: 10.1016/s0161-6420(98)92743-9. PMID 9479279
- [Background] Mori S, Hangai M, Sakamoto A, Yoshimura N. Spectral-domain optical coherence tomography measurement of macular volume for diagnosing glaucoma. J Glaucoma. 2010 Oct-Nov;19(8):528-34. doi: 10.1097/IJG.0b013e3181ca7acf. PMID 20164794
- [Background] Seong M, Sung KR, Choi EH, Kang SY, Cho JW, Um TW, Kim YJ, Park SB, Hong HE, Kook MS. Macular and peripapillary retinal nerve fiber layer measurements by spectral domain optical coherence tomography in normal-tension glaucoma. Invest Ophthalmol Vis Sci. 2010 Mar;51(3):1446-52. doi: 10.1167/iovs.09-4258. Epub 2009 Oct 15. PMID 19834029
- [Background] Kim NR, Lee ES, Seong GJ, Kim JH, An HG, Kim CY. Structure-function relationship and diagnostic value of macular ganglion cell complex measurement using Fourier-domain OCT in glaucoma. Invest Ophthalmol Vis Sci. 2010 Sep;51(9):4646-51. doi: 10.1167/iovs.09-5053. Epub 2010 Apr 30. PMID 20435603
- [Background] Hodapp E, Parrish RK II, Anderson DR. Clinical Decisions in Glaucoma. St. Louis, MO: Mosby; 1993:52- 61
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132